CLINICAL TRIAL: NCT05355454
Title: A Multicenter, Prospective, Randomized Controlled Clinical Study of STYLAGE® XXL Versus No-Treatment for Volume Deficiency in the Mid-face
Brief Title: Study of STYLAGE® XXL for Volume Deficiency in the Mid-Face
Acronym: MidFaceXXL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laboratoires Vivacy (Industry)
Collaborators: Avania B.V. (Unknown); Canfield Scientific Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VIV-STYL-XXL-02
Record Dates: First submitted 2022-04-25; First posted 2022-05-02 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Volume Deficiency in the Mid-Face; Aging; Aesthetics
Keywords: Mid-Face; Hyaluronic Acid; Volume; Aging; Aesthetics

STUDY DESIGN:
Intervention Model Description: Multi-Center, Prospective, Randomized, No-Treatment Controlled Trial. Subjects will be randomized (5:1 ratio) to the STYLAGE® XXL (treatment) arm or the no-treatment control arm.
  After 24 weeks, the no-treatment control arm (delayed treatment group) will receive their first treatment and will then follow the same schedule as the initial treatment group. After the no-treatment control group receives treatment, data from both groups will be pooled.
Who Masked: Outcomes Assessor
Masking Description: The primary endpoint is assessed through objective measures of facial volume, obtained using standardized, three-dimensional (3D), digital photographic images. Measurement will be made by an independent expert who will be blinded, as image files will not reveal subject treatment randomization, or the time point at which the image was taken.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STYLAGE® XXL Treatment Group (Experimental): Subjects randomized (5:1 ratio) to receive an initial treatment with STYLAGE® XXL Crosslinked Hyaluronic Acid Gel up to 8mL, based on the PI's assessment, in combination with the aesthetic goal of the subject, then an optional touch-up treatment session 4 weeks later, up to 4mL.
  Subjects will also be offered an optional retreatment at week 72 after initial treatment, up to 8mL.
  Interventions: Device: STYLAGE® XXL
- No-Treatment Control Group, then Delayed Treatment with STYLAGE® XXL (Other): No-Treatment for the first 6-month, then subjects will receive a delayed treatment with STYLAGE® XXL Crosslinked Hyaluronic Acid Gel up to 8mL, based on the PI's assessment, in combination with the aesthetic goal of the subject, then an optional touch-up treatment session 4 weeks later, up to 4mL.
  Subjects will also be offered an optional retreatment at week 72 after initial treatment, up to 8mL.
  Interventions: Device: STYLAGE® XXL

INTERVENTIONS:
Device: STYLAGE® XXL — Up to 2.0 mL will be injected in the zygomaticomalar region and optionally up to 2.0 mL in the anteromedial cheek at the first session, on each side of the face.
  Up to 1.0 mL in the zygomaticomalar region and optionally up to 1.0 mL in the anteromedial cheek for the optional touch-up session, on each side of the face.
  Up to 2.0 mL will be injected in the zygomaticomalar region and optionally up to 2.0 mL in the anteromedial cheek before study exit, on each side of the face.
  Arms: STYLAGE® XXL Treatment Group
Device: STYLAGE® XXL — Up to 2.0 mL will be injected in the zygomaticomalar region and optionally up to 2.0 mL in the anteromedial cheek at the first session, on each side of the face.
  Up to 1.0 mL in the zygomaticomalar region and optionally up to 1.0 mL in the anteromedial cheek for the optional touch-up session, on each side of the face.
  Up to 2.0 mL will be injected in the zygomaticomalar region and optionally up to 2.0 mL in the anteromedial cheek before study exit, on each side of the face.
  Arms: No-Treatment Control Group, then Delayed Treatment with STYLAGE® XXL

SUMMARY:
The primary objective of the study is to demonstrate the superiority of STYLAGE® XXL versus no treatment at 24 weeks after baseline for the creation or restoration of volume deficit in the mid-face.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, no-treatment controlled post-market clinical follow-up of a class III medical device. This study is designed to evaluate the safety and effectiveness of STYLAGE® XXL in the restorationor creation of volume in the mid-face.

The objective of this study is to demonstrate the superiority of STYLAGE® XXL versus no treatment at 24 weeks after baseline for the creation or restoration of volume deficit in the mid-face.

Assessment of superiority will be based on 3D analysis of the volumetric change, using a validated imaging system.

Effectiveness of STYLAGE® XXL will be demonstrated if the mean volumetric change at 24 weeks after baseline from pre-treatment in the treatment group is statistically superior to the mean change in the delayed treatment (control) group.

In total, approximately 90 subjects will be enrolled across three study centers in Switzerland, Austria, and France.

Subjects will be randomized to the treatment group or delayed treatment (control) group at a 5:1 ratio (i.e., there will be 5 more subjects treated with STYLAGE® XXL at baseline as compared to subjects who will be in the no-treatment (control) group and who will receive a delayed treatment with STYLAGE® XXL at 24 weeks after baseline).

The total duration of subject participation ranges from 18-19 months (treatment group) to 24-25 months (delayed treatment (control) group). Overall study duration including the enrolment period is expected to take approximately 30-31 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 30 and 65 years
* Seeking correction of his/her mid-face volume deficit, and agrees with recommendation by the Investigator
* Accept the obligation not to receive any other facial procedures or treatments impacting facial volume augmentation at any time during the study
* Able to follow study instructions and likely to complete all required visits, as assessed by the Investigator
* Psychologically able to understand the study related information and to give a written informed consent
* Have voluntarily provided written informed consent to participate in the study, and use of data privacy (sign the ethics committee approved Informed Consent Form), prior to any study-related procedure being performed
* Female of childbearing potential (sexually active, not sterile, nor postmenopausal for at least 1 year) must have a negative urine pregnancy test (UPT) at Visit 1 (or Visit 1b), and use a medically accepted contraceptive regimen since at least 12 weeks before the beginning of the study and for the duration of the study
* Affiliated to a health social security system (for France only)

Exclusion Criteria:

In terms of population:

* Pregnant or breastfeeding woman, or planning a pregnancy during the study
* Scars, moles, tattoo, or anything on the face which might interfere with the evaluation
* Subject who had been deprived of their freedom by administrative or legal decision or who is under guardianship
* Subject in a social or sanitary establishment
* Subject participating to another research on human beings or who is in an exclusion period of one
* Subject having received 4500 euros indemnities for participation in researches involving human beings in the 12 previous months, including participation in the present study (for France only)

In terms of associated pathology:

* Subject presenting any symptom which can be related to a medical condition that is likely to make the subject not being compliant with the study schedule, at the discretion of the investigator
* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results
* Subject with known history of or suffering from autoimmune disease and/or immune deficiency
* Subject suffering from active inflammatory and/or infectious cutaneous disorders in or near the studied zones (e.g. herpes, acne). Subject with recurrent herpes in the Midface area is not eligible even if asymptomatic at time of inclusion
* Subject prone to develop inflammatory skin conditions or having tendency to bleeding disorders
* Subject having history of allergy or anaphylactic shock including hypersensitivity to hyaluronic acid or to one of the components of the tested device
* Subject with a history of streptococcal disease, such as acute rheumatic fever or recurrent sore throats with cardiac localisation
* Subject with a tendency to develop keloids or hypertrophic scars

Relating to previous or ongoing treatment:

* Subject having received treatment with a laser, a dermabrasion, a surgery, a peeling, or other ablative procedure on the Midface area within the past 12 months prior to inclusion
* Subject having received injection with a resorbable filling product in the Midface area within the past 18 months prior to inclusion
* Subject having received at any time injection with a slowly resorbable filling product (e.g. polylactic acid, calcium hydroxyapatite, combinations of HA and Hypromellose) or with a non-resorbable filling product (e.g. polyacrylamide or silicone)
* Subject having received at any time a treatment with tensor threads in the Midface area
* Subject under medications which may cause lipo-atrophy
* Subject using medication such as aspirin, NSAIDs (e.g. ibuprofen), antiplatelet agents, anticoagulants, vitamin C within one week prior to inclusion and not agreeing not to take such treatments within 1 week prior to visit 2 (M1) or being a chronic user of anticoagulant treatment
* Subject undergoing a topical treatment on the test area or a systemic treatment:
* Antihistamines during the 2 weeks prior to study start
* Immunosuppressors and/or corticoids during the 4 weeks prior to study start
* Retinoids during the 6 months prior to study start

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Mid-Face Volumetric change | 24 weeks after baseline
  Mean volumetric change between the treatment group and no-treatment control group at 24 (V4) weeks after baseline (V1)

SECONDARY OUTCOMES:
Mid-Face Volumetric change | 4, and 12 weeks after baseline
  Mean volumetric change between the treatment group and no-treatment control group at 4 (V2) and 12 (V3) weeks after baseline (V1)
Mid-Face Volumetric change | 4, 12, 24, 48, and 72 weeks after initial treatment
  Mean volumetric change between pre-treatment and directly after treatment at V1 (or V1b), and 4 (V2/V2b), 12 (V3/V3b), 48 (V5), and 72 (V6) weeks after initial treatment, in both groups pooled.
Global Aesthetic Improvement, by the Subjects | 4, 12, and 24 weeks after baseline
  Global Aesthetic Improvement Scale (GAIS; improvement in the mid-face Area), assessed by the Subjects, between the treatment group and no-treatment control group.
  GAIS (Global Aesthetic Improvement Scale) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, with higher scores mean better improvement, with 1 means "Worse" and 5 means "Very much improved".
Global Aesthetic Improvement, by the Subjects | 4, 12, 24, 48, and 72 weeks after initial treatment
  Global Aesthetic Improvement Scale (GAIS; improvement in the mid-face Area), assessed by the Subjects, in both groups pooled.
  GAIS (Global Aesthetic Improvement Scale) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, with higher scores mean better improvement, with 1 means "Worse" and 5 means "Very much improved".
Global Aesthetic Improvement, by the Investigators | 4, 12, and 24 weeks after baseline
  Global Aesthetic Improvement Scale (GAIS; improvement in the mid-face Area), assessed by the Investigators, between the treatment group and no-treatment control group.
  GAIS (Global Aesthetic Improvement Scale) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, with higher scores mean better improvement, with 1 means "Worse" and 5 means "Very much improved".
Global Aesthetic Improvement, by the Investigators | 4, 12, 24, 48, and 72 weeks after initial treatment
  Global Aesthetic Improvement Scale (GAIS; improvement in the mid-face Area), assessed by the Investigators, in both groups pooled.
  GAIS (Global Aesthetic Improvement Scale) is a 5-point scale rating global aesthetic improvement in appearance, compared to pretreatment, with higher scores mean better improvement, with 1 means "Worse" and 5 means "Very much improved".
FACE-Q, by the Subjects | Baseline, and 4, 12, and 24 weeks after baseline
  Rash-transformed score of the FACE-Q, assessed by the Subjects, between the treatment group and no-treatment control group.
  FACE-Q is a patient-reported outcome (PRO) measure that can be used to measure outcomes of aesthetic facial procedures and products from the patient's perspective, composed of a set of independently functioning scales/checklists. In this study; two scales are assessed:
  1. FACE-Q - Satisfaction with cheekbones: This questionnaire consists of 10 items, and measures the appearance of cheekbones with items that ask about shape, contour and symmetry, as well as how attractive, high and well-defined the cheekbones look.
  2. FACE-Q - Satisfaction with outcome. This questionnaire consists of 6 items, and measures satisfaction with the result of a facial procedure, e.g., pleased with the result, result is fantastic.
  The total score is converted to a score from 0 to 100, with higher scores reflect a better outcome.
FACE-Q, by the Subjects | Initial treatment, and 4, 12, 24, 48, and 72 weeks after initial treatment
  Rash-transformed score of the FACE-Q, assessed by the Subjects, in both groups pooled.
  FACE-Q is a patient-reported outcome (PRO) measure that can be used to measure outcomes of aesthetic facial procedures and products from the patient's perspective, composed of a set of independently functioning scales/checklists. In this study; two scales are assessed:
  1. FACE-Q - Satisfaction with cheekbones: This questionnaire consists of 10 items, and measures the appearance of cheekbones with items that ask about shape, contour and symmetry, as well as how attractive, high and well-defined the cheekbones look.
  2. FACE-Q - Satisfaction with outcome. This questionnaire consists of 6 items, and measures satisfaction with the result of a facial procedure, e.g., pleased with the result, result is fantastic.
  The total score is converted to a score from 0 to 100, with higher scores reflect a better outcome.
Wrinkle Severity Rating Scale (WSRS), by the Investigators. | 4, 12, and 24 weeks after baseline
  Nasolabial Fold Severity using the wrinkle severity rating scale (WSRS), assessed by the Investigators, between the treatment group and no-treatment control group.
  The WSRS (Wrinkle Severity Rating Scale) is a 5-point rating scale to determine the severity of the nasolabial folds (NLF), with lower scores mean better condition (less severity), with 1 means "Absent - No visible NLF, continuous skin line" and 5 means "Extreme - Extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched".
Wrinkle Severity Rating Scale (WSRS), by the Investigators. | 4, 12, 24, 48, and 72 weeks after initial treatment
  Nasolabial Fold Severity using the wrinkle severity rating scale (WSRS), assessed by the Investigators, in both groups pooled.
  The WSRS (Wrinkle Severity Rating Scale) is a 5-point rating scale to determine the severity of the nasolabial folds (NLF), with lower scores mean better condition (less severity), with 1 means "Absent - No visible NLF, continuous skin line" and 5 means "Extreme - Extremely deep and long nasolabial fold, detrimental to facial appearance; 2-4 mm visible V-shaped fold when stretched".
Ease of sculpting and massaging, by the Investigators | Initial treatment, and 4, and 72 weeks after initial treatment
  Ease of sculpting and massaging of the HA gel, assessed by the investigator after each treatment session, on a 5-point scale ranging from "Very easy" to "Very difficult", in both groups pooled.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé RASPALDO, MD, Principal Investigator — Private Clinic, GENEVA, SWITZERLAND; Hugues CARTIER, MD, Principal Investigator — Centre Medical Saint-Jean, ARRAS, FRANCE; Thomas RAPPL, MD, Principal Investigator — Medical Aesthetic Research Academy, GRAZ, AUSTRIA; Cyril CLERICO, MD, Principal Investigator — Private Practice, NICE, FRANCE
Locations (1):
- Centre Medical Saint Jean, Arras, France

IPD SHARING:
Plan to Share IPD: No